CLINICAL TRIAL: NCT00953147
Title: A 6-Month Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Efficacy and Safety Study of Once Daily Ciclesonide HFA Nasal Aerosol (80 and 160 μg) in The Treatment of Perennial Allergic Rhinitis (PAR) in Subjects 12 Years and Older
Brief Title: A 6 Month Safety and Efficacy Study of Once Daily Ciclesonide Hydrofluoroalkane (HFA) in the Treatment of Perennial Allergic Rhinitis (PAR) in Subjects 12 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060-633
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Allergic Rhinitis; Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ciclesonide HFA 80 mcg once daily (Experimental): Ciclesonide HFA nasal aerosol will be supplied in a 40 mcg canister, to be administered as 1 puff in each nostril (80 mcg per day).
  Interventions: Drug: Ciclesonide HFA 80 mcg
- Ciclesonide HFA 160 mcg once daily (Experimental): Ciclesonide HFA nasal aerosol will be supplied in a 80 mcg canister, to be administered as 1 puff in each nostril (160 mcg per day).
  Interventions: Drug: Ciclesonide HFA 160 mcg
- Placebo once daily (Placebo Comparator): The placebo HFA nasal aerosol is identical to active drug, but does not contain ciclesonide.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide HFA 80 mcg — Ciclesonide HFA Nasal Aerosol 80 mcg once daily for 6 months in the treatment of Perennial Allergic Rhinitis (PAR) in subjects 12 years and older.
  Arms: Ciclesonide HFA 80 mcg once daily
Drug: Ciclesonide HFA 160 mcg — Ciclesonide HFA Nasal Aerosol 160 mcg once daily for 6 months in the treatment of Perennial Allergic Rhinitis (PAR) in subjects 12 years and older.
  Arms: Ciclesonide HFA 160 mcg once daily
Drug: Placebo — Placebo HFA Nasal Aerosol once daily for 6 months in the treatment of Perennial Allergic Rhinitis (PAR) in subjects 12 years and older.
  Arms: Placebo once daily

SUMMARY:
This is a 6-month multi-center, randomized, double-blind, placebo-controlled, parallel group, efficacy and safety study of ciclesonide HFA nasal aerosol administered once-daily to male and female subjects 12 years or older diagnosed with perennial allergic rhinitis (PAR).

DETAILED DESCRIPTION:
This study will investigate the efficacy and safety of once daily ciclesonide HFA Nasal Aerosol for 26 weeks. The primary objective is to evaluate the efficacy of ciclesonide HFA (80 mcg and 160 mcg) over 6 weeks, compared to placebo in subjects with PAR. Secondary objectives are to evaluate safety and tolerability and quality of life after treatment with ciclesonide HFA (80 mcg and 160 mcg), over 6 weeks and over 6 months.

The study will consist of a Screening period (7 to 21 (±3) days) from Visit 1 to Visit 2, followed by a Single-blind Placebo Run-in period (7 to 10 days) from Visit 2 to Visit 3, followed by a 6-month (26 weeks) double-blind treatment period (Visit 3 through Visit 11). Subjects who complete this study will be allowed to participate in a 6-month open-label extension study (Study 060-635).

This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent and assent, including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Subject must be in general good health based on screening physical examination, medical history, and clinical laboratory values.
* If any of the Screening visit Hematology, Chemistries, or Urinalysis are not within the clinical laboratory's reference range, then the subject can be included only if the Investigator judges the deviations to be not clinically significant.
* A history of PAR to a relevant perennial allergen (house dust mites, cockroach, molds, animal dander) for a minimum of two years immediately preceding the study Screening visit. The PAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past and require treatment throughout the entire study period.
* A demonstrated sensitivity at the Screening visit to at least one allergen known to induce PAR (house dust mite, animal dander, cockroach, and molds) using a standard skin-prick test. The subject's positive allergen test must be consistent with the medical history of PAR and must be present in the subject's environment throughout the study.
* Based upon subject's medical history, in the Investigator's judgment, the subject is unlikely to have a seasonal exacerbation during the first 6 weeks of double-blind treatment.
* Subject, if female ≤65 years of age, must have a negative serum pregnancy test at screening. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations; recent nasal biopsy; nasal trauma; or nasal ulcers or perforations. Surgery and atrophic rhinitis or rhinitis medicamentosa are not permitted within the last 60 days prior to the Screening visit.
* Subject is, in the investigator's judgement, having a seasonal exacerbation at the time of screening.
* Participation in any investigational drug trial within the 30 days preceding the Screening visit or planned participation in another investigational drug trial at any time during this trial.
* A known hypersensitivity to any corticosteroid or any of the excipients in the formulation of ciclesonide.
* History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, influenza, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening visit.
* History of alcohol or drug abuse within 2 years preceding the Screening visit .
* History of a positive test for HIV, hepatitis B or hepatitis C.
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta agonists and any controller drugs (eg, theophylline, leukotriene antagonists, etc.); intermittent use (less than or equal to 3 uses per week) of inhaled short acting beta-agonists is acceptable. Use of short acting beta-agonists for exercise-induced bronchospasm will be allowed.
* Expected use of any disallowed concomitant medications during the treatment period.
* Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit and use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
* Previous participation in an intranasal ciclesonide HFA nasal aerosol study.
* Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit.
* Initiation of pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or planned dose escalation during the study period.
* Study participation by clinical investigator site employees and/or their immediate relatives who reside in the same household.
* Study participation by more than one subject from the same household.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial:

  * impaired hepatic function including alcohol related liver disease or cirrhosis
  * history of ocular disturbances, eg, glaucoma or posterior subcapsular cataracts
  * any systemic infection
  * hematological, hepatic, renal, endocrine (except for controlled diabetes mellitus or postmenopausal symptoms or hypothyroidism)
  * gastrointestinal disease
  * malignancy (excluding basal cell carcinoma)
  * current neuropsychological condition with or without drug therapy • Any condition that, in the judgment of the investigator, would preclude the subject from completing the protocol with capture of the assessments as written.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1110 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Asthma and Allergy Specialists Medical Group, Huntington Beach, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - CHOC PSF, AMC, Division of Allergy Asthma & Immunology, Orange, California
  - California Allerga and Asthma Medical Group, Palmdale, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Bensch Research Associates, Stockton, California
  - Asthma and Allergy Associates, P.C., Colorado Springs, Colorado
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, Denver, Colorado
  - Clinical Research Atlanta, Atlanta, Georgia
  - DataQuest Medical Research, LLC, Lawrenceville, Georgia
  - Allergy and Asthma Consultants, PC, Lilburn, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Clinical Research Center of Indiana, Indianapolis, Indiana
  - Gordon D. Raphael, MD, Bethesda, Maryland
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Clinical Research Group of Montana, Bozeman, Montana
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Allergy and Asthma Center of NC, High Point, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Baker Allergy, Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Valley Clinical Research Center, Bethlehem, Pennsylvania
  - Asthma and Allergy Research Associates, Upland, Pennsylvania
  - Asthma, Nasal Disease and Allergy Research Center of New England, Providence, Rhode Island
  - National Allergy, Asthma, and Urticaria, Charleston, South Carolina
  - Allergy and Asthma Associates, Austin, Texas
  - Sirius Clinical Research, Austin, Texas
  - Hill Country Family Medical Center, Boerne, Texas
  - Pharmaceutical Research and Consulting, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - North Texas Institute for Clinical Trials, Fort Worth, Texas
  - Allergy and Asthma Associates, Houston, Texas
  - Kerrville Research Associates, PA, Kerrville, Texas
  - Kerrville Research Associates, Kerrville, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Southwest Allergy and Asthma Center, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - ASTHMA, Inc., Seattle, Washington

REFERENCES:
- [Result] Mohar D, Berger WE, Laforce C, Raphael G, Desai SY, Huang H, Hinkle J. Efficacy and tolerability study of ciclesonide nasal aerosol in patients with perennial allergic rhinitis. Allergy Asthma Proc. 2012 Jan-Feb;33(1):19-26. doi: 10.2500/aap.2012.33.3522. PMID 22370530

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Started | 298 | 505 | 307
Completed | 261 | 439 | 265
Not Completed | 37 | 66 | 42
Not completed — Adverse Event | 8 | 16 | 6
Not completed — Protocol Violation | 2 | 8 | 4
Not completed — Withdrawal by Subject | 13 | 15 | 12
Not completed — Lost to Follow-up | 8 | 9 | 4
Not completed — Physician Decision | 2 | 7 | 3
Not completed — Other | 4 | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily | Total
Number analyzed (Participants) | 298 | 505 | 307 | 1110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 44 | 17 | 88
  Between 18 and 65 years | 264 | 455 | 282 | 1001
  >=65 years | 7 | 6 | 8 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 37.5 (14.3) | 36.5 (13.2) | 38.0 (13.1) | 37.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 310 | 210 | 716
  Male | 102 | 195 | 97 | 394
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 94 | 60 | 216
  Not Hispanic or Latino | 236 | 411 | 247 | 894
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity [Number; unit: participants]
  White/Caucasian | 249 | 420 | 253 | 922
  Black or African American | 40 | 65 | 41 | 146
  Asian | 3 | 5 | 10 | 18
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 4 | 0 | 4
  Other | 3 | 6 | 3 | 12
  Multiple | 1 | 5 | 0 | 6
Baseline Reflective Total Nasal Symptom Score (rTNSS) [Mean (Standard Deviation); unit: units on a scale] — TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale
    AM | 8.51 (1.89) | 8.48 (1.88) | 8.60 (1.96) | 8.52 (1.90)
    PM | 8.53 (1.91) | 8.54 (1.84) | 8.64 (1.92) | 8.57 (1.88)
    AM and PM | 8.53 (1.82) | 8.50 (1.81) | 8.62 (1.88) | 8.54 (1.83)
Baseline Instanteous Total Nasal Symptom Score (iTNSS) [Mean (Standard Deviation); unit: units on a scale] — TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale
    AM | 7.93 (2.27) | 7.89 (2.24) | 8.01 (2.37) | 7.93 (2.29)
    PM | 7.38 (2.43) | 7.38 (2.41) | 7.39 (2.55) | 7.38 (2.46)
    AM and PM | 7.66 (2.28) | 7.64 (2.27) | 7.70 (2.38) | 7.66 (2.30)
Baseline Reflective Nasal Symptom Score (rNSS) [Mean (Standard Deviation); unit: units on a scale] — NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Reflective NSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale
    AM Sneezing | 1.73 (0.73) | 1.71 (0.72) | 1.75 (0.74) | 1.73 (0.73)
    AM Runny Nose | 2.24 (0.59) | 2.22 (0.59) | 2.28 (0.60) | 2.24 (0.59)
    AM Nasal Itching | 2.06 (0.64) | 2.08 (0.62) | 2.09 (0.69) | 2.08 (0.64)
    AM Nasal Congestion | 2.48 (0.49) | 2.46 (0.49) | 2.47 (0.53) | 2.47 (0.50)
    PM Sneezing | 1.81 (0.68) | 1.81 (0.70) | 1.88 (0.69) | 1.83 (0.69)
    PM Runny Nose | 2.23 (0.59) | 2.23 (0.60) | 2.27 (0.60) | 2.24 (0.60)
    PM Nasal Itching | 2.08 (0.64) | 2.12 (0.60) | 2.12 (0.69) | 2.11 (0.64)
    PM Nasal Congestion | 2.42 (0.53) | 2.38 (0.52) | 2.38 (0.54) | 2.39 (0.53)
    AM and PM Sneezing | 1.77 (0.68) | 1.76 (0.69) | 1.81 (0.69) | 1.78 (0.69)
    AM and PM Runny Nose | 2.24 (0.56) | 2.22 (0.58) | 2.27 (0.58) | 2.24 (0.57)
    AM and PM Nasal Itching | 2.07 (0.62) | 2.10 (0.60) | 2.11 (0.67) | 2.09 (0.62)
    AM and PM Nasal Congestion | 2.45 (0.48) | 2.42 (0.48) | 2.42 (0.51) | 2.43 (0.49)
Baseline Instantaneous Nasal Symptom Score (iNSS) [Mean (Standard Deviation); unit: units on a scale] — NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent (no sign/symptom evident);
  1. = mild
  2. = moderate
  3. = severe Instantaneous NSS measures these symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale
    AM Sneezing | 1.38 (0.91) | 1.40 (0.88) | 1.43 (0.93) | 1.40 (0.91)
    AM Runny Nose | 2.14 (0.68) | 2.13 (0.68) | 2.20 (0.67) | 2.15 (0.68)
    AM Nasal Itching | 2.00 (0.72) | 1.99 (0.69) | 2.00 (0.76) | 2.00 (0.72)
    AM Nasal Congestion | 2.41 (0.53) | 2.38 (0.56) | 2.38 (0.60) | 2.39 (0.57)
    PM Sneezing | 1.30 (0.90) | 1.32 (0.89) | 1.36 (0.90) | 1.32 (0.90)
    PM Runny Nose | 1.98 (0.73) | 1.98 (0.74) | 2.02 (0.72) | 1.99 (0.73)
    PM Nasal Itching | 1.87 (0.73) | 1.90 (0.71) | 1.83 (0.80) | 1.87 (0.74)
    PM Nasal Congestion | 2.22 (0.61) | 2.19 (0.63) | 2.17 (0.66) | 2.19 (0.63)
    AM and PM Sneezing | 1.35 (0.89) | 1.36 (0.86) | 1.39 (0.89) | 1.36 (0.88)
    AM and PM Runny Nose | 2.06 (0.67) | 2.05 (0.68) | 2.11 (0.65) | 2.07 (0.67)
    AM and PM Nasal Itching | 1.94 (0.70) | 1.95 (0.68) | 1.91 (0.75) | 1.93 (0.70)
    AM and PM Nasal Congestion | 2.32 (0.54) | 2.28 (0.57) | 2.28 (0.60) | 2.29 (0.57)
Baseline Rhinoconjunctivitis Quality of Life Questionnaire score [RQLQ (S)] )≥3.0 [Mean (Standard Deviation); unit: units on a scale] — Baseline Rhinoconjunctivitis Quality of Life Questionnaire [RQLQ(S)] Score in Subjects with baseline RQLQ(S) ≥3.0. RQLQ(s)consists of 28 questions, each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Domains: Activities (questions 1-3), Sleep (questions 4-6), Non-Nose/Eye Symptoms (questions 7-13), Practical Problems (questions 14-16), Nasal Symptoms (questions 17-20), Eye Symptoms (questions 21-24), and Emotional (questions 25-28). The overall RQLQ(S) score was calculated as the average of the mean domain scores.
  units on a scale | 4.16 (0.77) | 4.05 (0.76) | 4.12 (0.78) | 4.10 (0.77)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Subject-reported AM and PM Reflective TNSS (rTNSS) Averaged Over the First 6 Weeks of Double-blind Treatment
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the six week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 298 | 504 | 305
units on a scale | -1.97 (0.13) | -1.82 (0.10) | -1.28 (0.13)
Statistical Analysis 1: Comparison: Ciclesonide HFA 80 Mcg Once Daily vs Placebo Once Daily; The null hypothesis is that there is no difference in primary outcome when compare active to placebo group. The alternative hypothesis is that there is a difference in primary outcome when compare active to placebo group. It was estimated that 200 subjects per group will provide at least 85% power to detect a difference between treatment groups of 0.7 in the change from baseline in iTNSS with a two-sided alpha level of 0.025; Test type: Superiority or Other; p < 0.0001, ANCOVA — The p-value from primary outcome was adjusted at alpha=0.025; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [0.35 to 1.04]
Statistical Analysis 2: Comparison: Ciclesonide HFA 160 Mcg Once Daily vs Placebo Once Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0005, ANCOVA — The p-value from primary outcome was adjusted at alpha=0.025; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [0.24 to 0.84]

2. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM Instantaneous TNSS (iTNSS) Averaged Over the First 6 Weeks of Double-blind Treatment
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the six week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 298 | 504 | 305
units on a scale | -1.77 (0.12) | -1.60 (0.10) | -1.18 (0.12)
Statistical Analysis 1: Comparison: Ciclesonide HFA 80 Mcg Once Daily vs Placebo Once Daily; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p = 0.0014, ANCOVA; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [0.25 to 0.92]
Statistical Analysis 2: Comparison: Ciclesonide HFA 160 Mcg Once Daily vs Placebo Once Daily; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p = 0.0122, ANCOVA; Median Difference (Final Values) = 0.42, 95% CI 2-sided [0.12 to 0.72]

3. Secondary Outcome: Change From Baseline in Daily Subject-reported AM rTNSS Averaged Over the First 6 Weeks of Double-blind Treatment.
Description: as for outcome 1
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 297 | 503 | 304
units on a scale | -1.94 (0.13) | -1.78 (0.10) | -1.25 (0.13)

4. Secondary Outcome: Change From Baseline in Daily Subject-reported PM rTNSS Averaged Over the First 6 Weeks of Double-blind Treatment.
Description: as for outcome 1
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 298 | 504 | 305
units on a scale | -2.01 (0.13) | -1.88 (0.10) | -1.32 (0.13)

5. Secondary Outcome: Change From Baseline in Daily Subject-reported AM iTNSS Averaged Over the First 6 Weeks of Double-blind Treatment.
Description: as for outcome 2
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all participants analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 297 | 503 | 304
units on a scale | -1.78 (0.12) | -1.67 (0.10) | -1.23 (0.12)

6. Secondary Outcome: Change From Baseline in Daily Subject-reported PM iTNSS Averaged Over the First 6 Weeks of Double-blind Treatment.
Description: as for outcome 2
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 298 | 504 | 305
units on a scale | -1.76 (0.13) | -1.55 (0.10) | -1.15 (0.13)

7. Secondary Outcome: Change From Baseline in Daily Subject-reported AM rNSS Averaged Over the First 6 Weeks of the Double-blind Treatment
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Reflective NSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the six week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0 - 6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 297 | 503 | 304
units on a scale
  Sneezing | -0.51 (0.04) | -0.47 (0.03) | -0.31 (0.04)
  Runny Nose | -0.49 (0.04) | -0.44 (0.03) | -0.31 (0.04)
  Nasal Itching | -0.52 (0.04) | -0.48 (0.03) | -0.38 (0.04)
  Nasal Congestion | -0.42 (0.03) | -0.38 (0.03) | -0.25 (0.03)

8. Secondary Outcome: Change From Baseline in Daily Subject-reported PM rNSS Averaged Over the First 6 Weeks of the Double-blind Treatment
Description: as for outcome 7
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 298 | 504 | 305
units on a scale
  Sneezing | -0.53 (0.04) | -0.52 (0.03) | -0.35 (0.04)
  Runny Nose | -0.51 (0.04) | -0.47 (0.03) | -0.31 (0.04)
  Nasal Itching | -0.54 (0.04) | -0.51 (0.03) | -0.39 (0.04)
  Nasal Congestion | -0.43 (0.03) | -0.39 (0.03) | -0.26 (0.03)

9. Secondary Outcome: Change From Baseline in Daily Subject-reported AM & PM rNSS Averaged Over the First 6 Weeks of Double-blind Treatment Period.
Description: as for outcome 7
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 298 | 504 | 305
units on a scale
  Sneezing | -0.52 (0.04) | -0.49 (0.03) | -0.33 (0.04)
  Runny Nose | -0.50 (0.04) | -0.45 (0.03) | -0.31 (0.04)
  Nasal Itching | -0.53 (0.04) | -0.49 (0.03) | -0.39 (0.04)
  Nasal Congestion | -0.42 (0.03) | -0.39 (0.03) | -0.26 (0.03)

10. Secondary Outcome: Change From Baseline in Daily Subject-reported AM iNSS Averaged the First 6 Weeks of the Double-blind Treatment
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Instantaneous NSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the six week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 297 | 503 | 304
units on a scale
  Sneezing | -0.45 (0.04) | -0.44 (0.03) | -0.34 (0.04)
  Runny Nose | -0.47 (0.04) | -0.43 (0.03) | -0.30 (0.04)
  Nasal Itching | -0.51 (0.04) | -0.47 (0.03) | -0.37 (0.04)
  Nasal Congestion | -0.36 (0.03) | -0.33 (0.02) | -0.22 (0.03)

11. Secondary Outcome: Change From Baseline in Daily Subject-reported PM iNSS Averaged the First 6 Weeks of the Double-blind Treatment
Description: as for outcome 10
Time Frame: Weeks 0-6
Population: Intent to Treat Population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 298 | 505 | 307
units on a scale
  Sneezing | -0.44 (0.04) | -0.39 (0.03) | -0.31 (0.04)
  Runny Nose | -0.47 (0.04) | -0.40 (0.03) | -0.29 (0.04)
  Nasal Itching | -0.49 (0.04) | -0.45 (0.03) | -0.33 (0.04)
  Nasal Congestion | -0.37 (0.03) | -0.31 (0.03) | -0.22 (0.03)

12. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM iNSS Averaged Over the First 6 Weeks of Double-blind Treatment Period
Description: as for outcome 10
Time Frame: Weeks 0-6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 298 | 504 | 305
units on a scale
  Sneezing | -0.44 (0.04) | -0.41 (0.03) | -0.32 (0.04)
  Runny Nose | -0.47 (0.04) | -0.41 (0.03) | -0.30 (0.04)
  Nasal Itching | -0.50 (0.04) | -0.46 (0.03) | -0.35 (0.04)
  Nasal Congestion | -0.36 (0.03) | -0.32 (0.02) | -0.22 (0.03)

13. Secondary Outcome: Change From Baseline to Week 6 in Rhinoconjunctivitis Quality of Life Questionnaire With Standardized [RQLQ(S)] Overall Score in Impaired Patients With Baseline RQLQ(S) Score ≥3.0
Description: RQLQ(S) scores in subjects with baseline RQLQ[S] score ≥3.0. RQLQ(S) consists of 28 questions, each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Domains: Activities (questions 1-3), Sleep (questions 4-6), Non-Nose/Eye Symptoms (questions 7-13), Practical Problems (questions 14-16), Nasal Symptoms (questions 17-20), Eye Symptoms (questions 21-24), and Emotional (questions 25-28). The overall RQLQ(S) score was calculated as the average of the mean domain scores.
Time Frame: Baseline and Week 6
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 109 | 191 | 101
units on a scale | -1.55 (0.13) | -1.27 (0.11) | -0.96 (0.14)

14. Secondary Outcome: Change From Baseline to Month 6 (Week 26) in RQLQ(S) Overall Score in Impaired Patients With Baseline RQLQ(S) Score ≥3.0.
Description: RQLQ(S) scores in impaired subjects with baseline RQLQ[S] score ≥3.0. RQLQ(S)consists of 28 questions, each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Domains: Activities (questions 1-3), Sleep (questions 4-6), Non-Nose/Eye Symptoms (questions 7-13), Practical Problems (questions 14-16), Nasal Symptoms (questions 17-20), Eye Symptoms (questions 21-24), and Emotional (questions 25-28). The overall RQLQ(S) score was calculated as the average of the mean domain scores.
Time Frame: Baseline and Week 26
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 100 | 160 | 86
units on a scale | -1.67 (0.14) | -1.62 (0.11) | -1.40 (0.15)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Ciclesonide HFA 80 Mcg Once Daily | Ciclesonide HFA 160 Mcg Once Daily | Placebo Once Daily
Serious Adverse Events (participants affected / at risk) | 6/298 | 8/505 | 6/307
Other Adverse Events (participants affected / at risk) | 148/334 | 234/475 | 131/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide HFA 80 Mcg Once Daily (N=298) | Ciclesonide HFA 160 Mcg Once Daily (N=505) | Placebo Once Daily (N=307)
Artrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic atony (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia obstructive (General disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mononeuropathy mulitplex (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Imprisonment (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide HFA 80 Mcg Once Daily (N=334) | Ciclesonide HFA 160 Mcg Once Daily (N=475) | Placebo Once Daily (N=243)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 7 (8) | 7 (7)
Nausea (Gastrointestinal disorders) | 9 (10) | 8 (8) | 2 (2)
Instillation site discomfort (General disorders) | 10 (11) | 9 (11) | 0 (0)
Bronchitis (Infections and infestations) | 7 (7) | 11 (11) | 6 (6)
Influenza (Infections and infestations) | 6 (6) | 9 (11) | 3 (4)
Nasopharyngitis (Infections and infestations) | 14 (17) | 30 (35) | 19 (26)
Pharyngitis streptococcal (Infections and infestations) | 7 (8) | 5 (5) | 5 (6)
Sinusitis (Infections and infestations) | 14 (16) | 27 (30) | 17 (18)
Upper respiratory tract infection (Infections and infestations) | 43 (54) | 66 (74) | 29 (37)
Urinary tract infection (Infections and infestations) | 13 (13) | 14 (16) | 9 (10)
Viral upper respiratory tract infection (Infections and infestations) | 15 (16) | 13 (14) | 7 (9)
Muscle strain (Injury, poisoning and procedural complications) | 6 (7) | 7 (9) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (12) | 11 (11) | 10 (12)
Headache (Nervous system disorders) | 21 (36) | 17 (27) | 14 (18)
Sinus headache (Nervous system disorders) | 6 (10) | 4 (7) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 19 (19) | 8 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 34 (57) | 57 (98) | 24 (42)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 16 (16) | 2 (2)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (14) | 2 (2)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 16 (21) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 20 (22) | 10 (11)
Hypertension (Vascular disorders) | 4 (4) | 7 (8) | 8 (8)

LIMITATIONS AND CAVEATS:
This study was not designed or powered for a comparison of the 80mcg dose with the 160mcg dose therefore no statistical comparisons were planned between the two active groups. Publication references to 74 and 148mcg are equivalent to 80 and 160mcg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other